CLINICAL TRIAL: NCT01841086
Title: A Randomized, Open-label, Single Dose, 3-Treatment, 3-Period Williams-Design to Assess the Pharmacokinetic Characteristics and Food Effect of Sarpogrelate HCl CR Tablets Compared With Sarpogrelate HCl IR Tablets in Healthy Male Subjects
Brief Title: Pharmacokinetics and Food Effect of Sarpogrelate HCl CR Formulation in Comparison to Immediate-release Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Korea United Pharm. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KUP-SPG3-101
Record Dates: First submitted 2013-04-21; First posted 2013-04-26 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Healthy

ARMS (2):
- Anplag (Active Comparator): Sarpogrelate HCl 300mg once a day or 100mg three times a day
  Interventions: Drug: Anplag; Drug: UI03SPG300CT
- UI03SPG300CT (Experimental): Sarpogrelate HCl 300mg once a day or 100mg three times a day
  Interventions: Drug: Anplag; Drug: UI03SPG300CT

INTERVENTIONS:
Drug: Anplag — Sarpogrelate HCl 300mg once a day or 100mg three times a day
  Other Names: UI03SPG300CT
Drug: UI03SPG300CT — Sarpogrelate HCl 300mg once a day or 100mg three times a day

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of sarpogrelate controlled-release formulation (CR) in comparison to immediate-release formulation (IR) and Food effect on the pharmacokinetics of sarpogrelate CR.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 55 years of healthy volunteers

Exclusion Criteria:

* Hypersensitivity Reaction about Sarpogrelate HCl or other antiplatelets

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Cmax | 24h
  Active Comparator : predose(0), 0.25, 0.5, 1, 1.5, 2, 3, 6(immediately before 2nd drug intake) , 6.25, 6.5, 7, 7.5, 8, 9, 12(immediately before 3rd drug intake), 12.5, 13, 13.5, 14, 15, 16, 24 hours post-dose Experimental : predose(0), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24 hours post-dose
AUCt | 24h
  Active Comparator : predose(0), 0.25, 0.5, 1, 1.5, 2, 3, 6(immediately before 2nd drug intake) , 6.25, 6.5, 7, 7.5, 8, 9,12(immediately before 3rd drug intake), 12.5, 13, 13.5, 14, 15, 16, 24 hours post-dose Experimental : predose(0), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24 hours post-dose

SECONDARY OUTCOMES:
tmax, t1/2 | 24h
  Active Comparator : predose(0), 0.25, 0.5, 1, 1.5, 2, 3, 6(immediately before 2nd drug intake) , 6.25, 6.5, 7, 7.5, 8, 9, 12(immediately before 3rd drug intake), 12.5, 13, 13.5, 14, 15, 16, 24 hours post-dose Experimental : predose(0), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24 hours post-dose
AUC0-∞ | 24h
  Active Comparator : predose(0), 0.25, 0.5, 1, 1.5, 2, 3, 6(immediately before 2nd drug intake) , 6.25, 6.5, 7, 7.5, 8, 9,12(immediately before 3rd drug intake), 12.5, 13, 13.5, 14, 15, 16, 24 hours post-dose Experimental : predose(0), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Wooseong Huh, M.D., Ph.D., Principal Investigator — Samsung Medical Center